CLINICAL TRIAL: NCT06546618
Title: Little Cigar and Cigarillo Warnings to Reduce Tobacco-Related Cancers and Disease - Eye Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 24-0841; R01CA240732 (NIH)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Use
Keywords: Text-only warning messages; LCC packages with flavor descriptors; pictorial warnings messages; LCC packages without flavor descriptors
MeSH Terms: conditions — Tobacco Use | interventions — Candy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LCC Package with pictorial warning and no flavor (Experimental): Participants will see a mock LCC package with pictorial warnings and no flavor descriptor.
  Interventions: Behavioral: pictorial warning and no flavor
- LCC Package with pictorial warning and 'sweet' flavor (Experimental): Participants will see a mock LCC package with pictorial warnings and a 'sweet' flavor descriptor.
  Interventions: Behavioral: pictorial warning and 'sweet' flavor
- LCC Package with text-only warning and no flavor (Experimental): Participants will see a mock LCC package with text-only warnings and no flavor descriptor.
  Interventions: Behavioral: text-only warning and no flavor
- LCC Package with text-only warning and 'sweet' flavor (Experimental): Participants will see a mock LCC package with text-only warnings and a 'sweet' flavor descriptor
  Interventions: Behavioral: text-only warning and 'sweet' flavor

INTERVENTIONS:
Behavioral: pictorial warning and no flavor — LCC Package with pictorial warning and no flavor
  Arms: LCC Package with pictorial warning and no flavor
Behavioral: pictorial warning and 'sweet' flavor — LCC Package with pictorial warning and 'sweet' flavor
  Arms: LCC Package with pictorial warning and 'sweet' flavor
Behavioral: text-only warning and no flavor — LCC Package with text-only warning and no flavor
  Arms: LCC Package with text-only warning and no flavor
Behavioral: text-only warning and 'sweet' flavor — LCC Package with text-only warning and 'sweet' flavor
  Arms: LCC Package with text-only warning and 'sweet' flavor

SUMMARY:
The goal of this research is to determine how removal of little cigar and cigarillo (LCC) flavor descriptors on packaging impacts attention and affective responses to LCC warnings. A study will be conducted using eye tracking, electrodermal activity (galvanic skin response), and survey measures of affect to measure participant responses to LCC packages varied by warning type (pictorial vs. text only) and flavor contents ('Sweet' flavor descriptor vs. no flavor descriptor).

DETAILED DESCRIPTION:
Over 4 million US adults regularly smoke cigars, which causes multiple cancers, including oral, esophageal, pancreatic, laryngeal, and lung cancer. Even smoking 1-2 cigars per day is associated with elevated cancer risk. Though cigarette consumption decreased 39% from 2000 to 2015, cigar consumption increased 85%. Of the three major types of cigars-large cigars, little cigars, and cigarillos-little cigars and cigarillos (LCC) are the most commonly used in the US. LCC use among adults has increased in part because LCCs are taxed at a lower rate than cigarettes, are subject to fewer regulations and marketing restrictions, can be purchased in small pack sizes, and are exempt from flavor bans that apply to cigarettes.

In May 2016, the Food and Drug Administration (FDA) required text-only warnings on LCC packs, rotating among six statements. Research on cigarettes suggests warnings on packs should have multiple rotating sets, contain images illustrating the negative health effects associated with LCC use, and be large. However, the evidence for cigarette warning labels cannot adequately inform implementation of improved LCC warnings for four reasons: 1) The currently mandated cigar warnings differ from existing cigarette warnings; 2) there is no evidence on the effectiveness of the currently mandated cigar warnings (i.e., behavioral intentions or outcomes) or evidence on efforts that might improve LCC warnings (i.e., images, larger warning size, removal of LCC flavor descriptors on packaging); 3) Courts have ruled that one type of effective tobacco warning (i.e., for cigarettes) cannot be used to justify other types of tobacco warnings, such as those for LCCs and 4) LCC users have different demographic and consumption profiles than cigarette users (i.e., LCC users include a higher proportion of young adults African Americans, and LCCs are used on fewer days per month, which should be taken into account when developing improved warnings.

Gaps exist in understanding how LCC policies, such as the removal of flavor descriptors on packaging, influence the impact of LCC warnings. This eye tracking and psychophysiology project will provide new data to fill these evidence gaps and advance general scientific knowledge about elements of tobacco warnings research.

During the study, Participants will see 12 LCC pack stimuli images presented in random order. 3 packs will feature pictorial LCC warnings and a "Sweet" flavor descriptor, and the same 3 warnings will be presented on packs without a flavor. The remaining 6 LCC packs will have 3 text-only warnings, with 3 images containing the "Sweet" flavor and 3 images without a flavor. We will measure attention to the warnings and attention to the flavor descriptors as well as electrodermal activity and affective responses for each of the 12 stimuli.

ELIGIBILITY:
Participants will be recruited through flyers, emails, and recruitment websites to identify potentially eligible participants local to our study location (Chapel Hill/Carrboro, NC)

Inclusion Criteria:

* Over 21 years old
* Pass quality/bot screening (will answer honestly, captcha, simple math question)
* Speak English
* Current every day or some day users of LCC products
* Able to come to an appointment in NC triangle area
* Do not have any eye conditions that prevent them from being eye tracked (e.g., glaucoma, lazy eye, bifocals)

Exclusion Criteria:

* Under 21 years old
* Do not speak English
* Unable to pass quality/bot screening
* Unable to come to an appointment
* Eye conditions that prevent eye tracking (e.g., glaucoma, lazy eye, bifocals)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Attention to warning areas of interest | Baseline
  Attention to warning areas of interest will be measured by dwell time to pre-defined areas of interest on the little cigars or cigarillos (LCCs) package. The total amount of time in iseconds that participants spend looking at warnings will be determined.
Attention to flavor area of interest | Baseline
  Attention to flavor area of interest will be measured by dwell time to pre-defined areas of interest on the little cigars or cigarillos (LCCs) package. The total amount of time inseconds that people spend looking at the area where the flavor of the LCC is shown will be determined.

SECONDARY OUTCOMES:
Electrodermal activity | Baseline
  Electrodermal activity indexes emotional arousal by sensing sweat on the hands, it will be measured using a Shimmer 3 galvanic skin response sensor placed on the non-dominant hand.Electrodermal activity is measured in units of microsiemens (µS), an increase in electrodermal activity indicates an increase in emotional arousal.
Affective response to warnings | Baseline
  Affective response to warnings will be measured using an adaptation of the Discrete Emotions Questionnaire. The affective responses questionnaire will include 12 different emotions (6 positive, 6 negative) to measure participant's emotional responses to the cigarillo packages. Participants will rate to what extent they experienced each emotion while viewing the LCC package on a scale of 1 to 7, where 1=not at all and 7=an extreme amount. Higher affective responses indicate stronger emotional reactions to the LCC package.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Adam O Goldstein, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials